CLINICAL TRIAL: NCT04747704
Title: Establishing Preliminary Efficacy of Three Principles Correctional Counseling in a Prison Sample
Brief Title: Three-Principles Approach for Incarcerated Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Sarah Bowen, Associate Professor, Pacific University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206211-5
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Psychological Distress; Recidivism
MeSH Terms: conditions — Recidivism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants receiving Three-Principles Counseling
  Interventions: Behavioral: Three Principles Counseling

INTERVENTIONS:
Behavioral: Three Principles Counseling — A 10-week insight-based program offered in prisons in a group setting for 2 hours each week. Approximately 15 - 20 adults or youth in custody participate at a time, led by two trained teachers. The curriculum is designed to teach an understanding of the mind and human experience for the purpose of reducing risk factors, uncovering resiliency and to promote emotional and psychological well-being for adults and youth in the criminal justice system. This is taught through a compilation of sessions that speak to the potential, ability and resilience inherent in every individual. Sessions include a mix of lessons, experiential learning, and group conversations.

SUMMARY:
The purpose of the study is to examine the feasibility, acceptability and preliminary efficacy of an acceptance-based, insight-oriented treatment approach for US incarcerated adults. Feasibility and acceptability will be assessed through attendance and retention throughout the intervention period. Primary outcomes include negative affect, psychological flexibility, emotion regulation, purpose in life, impulsivity, and trauma. Changes will be assessed from baseline to post-course, post-course to 6-month follow up, and baseline to 6-month follow up for all primary outcomes. Researchers hypothesize that, 1) retention rates will be similar to previous trials with 70% retention from pre- to post-course; 2) there will be significant baseline-to-post-course reductions in psychological symptoms, impulsivity, and trauma, and an increase in psychological flexibility, purpose in life, and emotion regulation; and 3) there will be significant baseline-to-6-month reductions in psychological symptoms, impulsivity, and trauma, and an increase in psychological flexibility, purpose in life, and emotion regulation.

DETAILED DESCRIPTION:
Prevailing correctional counseling methods (e.g., cognitive-behavior therapy, social learning) often operate from an "outside-in" paradigm attempting to put mental health "into" people in prison using various strategies and techniques. Three Principles Correctional Counseling (3PCC), informed by theosophy of Sydney Banks, with a subsequent intervention based on Banks's work, is grounded in a different paradigm-in which all individuals, including incarcerated, have innate positive mental health; however, their belief systems convince them otherwise. When incarcerated individuals learn to navigate daily challenges with mental clarity, affective states shift from negative to positive, allowing for state-dependent positive recall, leading to lower likelihood of responding to negative thoughts and feelings with deviant and other health-damaging behavior.

Studies suggest 3PCC leads to improvements in negative affect such as depression, anxiety, and rumination, and increases in positive outcomes including mindfulness, mental health, social well-being, emotional regulation and non-attachment in non-correctional samples, reductions in stress and anxiety for HIV-positive patients; improvements in substance use problems, criminal justice involvement, employment, housing, and psychological wellbeing for women in in-patient substance abuse treatment; improved resilience in high-risk children and adolescents, improved mental health and resilience in young trauma-exposed sex offenders, improvements in thought recognition, mindfulness, and psychological well-being in a correctional sample, and improved in mental well-being, purpose in life, anxiety and anger, and behavior in a UK prison. 3PCC has also shown feasibility and acceptability in refugee women with trauma, and demonstrated feasible retention rates of 76% in an English prison setting.

The current trial is designed to further assess efficacy of 3PCC in incarcerated individuals. 3PCC classes will be facilitated by practitioners with several years of experience working with diverse client populations. Each 3PCC class will meet weekly for 10 consecutive weeks, with each session approximately 3 hours long. Classes will include the following modules: Building Rapport, Exploration of "Reality"; Separate Realities; Exploration of Thought and Insight; Consciousness-Where Does it Come From?; Exploring Feelings/Moods/Behavior; Exploring Innate Health/Natural Intelligence; What is Mind?; Exploring Infinite Potential; Exploring Mental Clarity Versus a Busy Mind; Stepping into the Unknown, Implications of the Principles for Life in Prison; and Living Outside of Prison.

Hypothesis 1: Compared with the control group, participants in the 3PCC condition will demonstrate significant increases in psychological flexibility, quality of life, clear mind, emotional regulation, impulse control and purpose in life at post-course, which will be maintained at 3- and 6-month follow-up.

Hypothesis 2: Compared with the control group, participants exposed to 3PCC will show significant decreases in depression, anxiety, anger, and trauma symptoms at post-course, which will be maintained at 3- and 6-month follow-up.

Hypothesis 3: Compared with the control group, participants exposed to 3PCC will show greater improvement in behavior within the prison community at post-course, which will be maintained at 3- and 6-month follow-up. Behavior will be measured by prison records measuring participants' behavioral violations and rewards for prosocial behavior.

ELIGIBILITY:
Inclusion Criteria:

* at least 9 months left in their sentence
* agree to complete assessments at baseline, post-course, and 3 and 6 months following completion of the 3PCC course
* are able to read and write in English.

Exclusion Criteria:

* DOC staff deems it inappropriate for them to participate in the study for clinical or administrative reasons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Flexibility and Experiential Avoidance across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The Acceptance and Action Questionnaire-II (Bond et al., 2011) is a self-report measure of experiential avoidance and psychological inflexibility.
Change in Wellbeing across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  Short Form 36 (SF-36) is a self-report measure assessing health-related quality of living.
Change in Emotion Regulation across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The DERS-18 is a brief, 18-item self-report questionnaire designed to assess multiple aspects of emotional dysregulation (Victor & Klonsky, 2016).
Change in Purpose in Life across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The PILT is a 20-item self-report attitude scale, which measures the extent to which people perceive their lives to be purposeful and meaningful.
Change in Trauma symptoms across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The PTSD Checklist - Civilian version (PCL-C; Weathers et al., 1994) is a 17-item self-report, diagnostic screening instrument assessing criteria for PTSD.
Change in Impulsivity across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking scale (UPPS; Whiteside & Lynam, 2001) is a self-report, 45-item inventory to measure four distinct personality pathways to impulsive behavior.
Change in Depression across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  PROMIS Depression-Short Form (PR-Dep; PROMIS Health Organization) is an 8-item self-report measure assessing depression based on DSM-5 symptomatology. Respondents report the degree to which they have been bothered by each symptom during the past 7 days.
Change in Anxiety across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The PROMIS Anxiety-Short Form (PR-Anx; PROMIS Health Organization) is a 7-item self-report measure assessing anxiety based on DSM-5 symptomatology. Respondents report the degree to which they have been bothered by each symptom during the past 7 days.
Change in Anger across 6 months | Pre-intervention, Post-intervention (10 weeks after Pre-intervention), 3 months and 6 months following Post-intervention
  The PROMIS Anger-Short Form (PR-Ang; PROMIS Health Organization) is a 5-item self-report scale measuring anger based on DSM-5 symptomatology. Respondents reported the degree to which they have been bothered by each symptom during the past 7 days.
Change in Prosocial and Non-Prosocial Behavior across 6 months | Pre-intervention, and 6 months following Post-intervention
  Prison records regarding participants' behavioral violations and rewards for pro-social behavior will provide data on prosocial and Non-Prosocial behaviors.

SECONDARY OUTCOMES:
Acceptability | Post-intervention (10 weeks after Pre-intervention)
  The Course Satisfaction Survey will be given out upon completion of the group (along with the post-intervention assessments) as a means of collecting qualitative data about what the participants felt they can take away from the group.

CONTACTS AND LOCATIONS:
Locations (1):
- Pcific University, Hillsboro, Oregon, United States